CLINICAL TRIAL: NCT04791943
Title: Preoperative Melatonin to Decrease Analgesia Usage After Third Molar Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Quest Diagnostics-Nichols Insitute (Industry); Eurofins Viracor (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-12127
Record Dates: First submitted 2021-03-02; First posted 2021-03-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Pain, Postoperative; Narcotic Use
MeSH Terms: conditions — Pain, Postoperative | interventions — Melatonin; Lactose

STUDY DESIGN:
Intervention Model Description: A randomization list using a variable block size will be prepared by the study biostatistician. The lists of treatment assignments (1:1 ratio) will be kept on file.
Who Masked: Participant, Care Provider
Masking Description: The surgeon and the patient will be masked, the research coordinator will not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Treatment - Melatonin (Experimental): Premedication for three nights with 10mg melatonin
  Interventions: Drug: Melatonin 10 MG
- Control Treatment - Lactose (Placebo Comparator): Premedication for three nights with lactose capsules
  Interventions: Drug: Lactose pill

INTERVENTIONS:
Drug: Melatonin 10 MG — 3 melatonin 10mg capsules will be given to the treatment arm
  Arms: Experimental Treatment - Melatonin
Drug: Lactose pill — 3 lactose pills will be provided to the control arm
  Arms: Control Treatment - Lactose

SUMMARY:
The purpose of the study is to assess if melatonin given for three nights before wisdom tooth surgery decreases post-operative pain and pain medication consumption. Patients will receive either melatonin or a placebo for three nights prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have 3-4 partial or full bony impacted third molars requiring surgical extraction under IV sedation
* Ages 18-35
* American Society of Anesthesiologists (ASA) Class I or II
* English or Spanish speaking patients
* Capacity to sign informed consent

Exclusion Criteria:

* Allergies to melatonin, opioids, or other Over-the-counter (OTC) pain medications
* Anyone currently taking melatonin for any reason
* Cases under local anesthesia
* ASA class III or higher
* Sleep disorder (insomnia/narcolepsy)
* Current or past history of substance abuse
* Chronic pain
* Language/communication barrier
* Psychiatric disease/ Mental impairment
* Current or past use of psychotropic drugs
* Pregnancy
* Renal or hepatic impairment
* BMI >35

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Postoperative narcotic consumption | From the time of intervention to the completion of the surveys, approximately 2-4 weeks total
  Postoperative consumption of narcotic pain medication will be measured for approximately 72 hours post operatively. Three total surveys will be administered. The surveys will be sent to participants via text message or email and include a link to SurveyMonkey. These surveys will be sent in the morning approximately 1 day, 2 days, and 3 days after surgery. The surveys will query for participant identification and then ask how many tablets of ibuprofen 600mg and hydrocodone-acetaminophen have been taken since the time of surgery or the time of previous survey depending on if the survey is received on Day 1, versus Day 2, and Day 3. The number of narcotic pain medication pills consumed postoperatively will be presented as means and standard deviations by treatment arm.

SECONDARY OUTCOMES:
Inflammatory cytokine markers - IL-6, IL-8, TNF-alpha concentrations | Blood draws during consultation, immediately prior to surgery, and at POD5, approximately 2-4 weeks total
  Preoperative and postoperative blood draws will be taken to measure concentrations of the inflammatory biomarkers Interleukin-6 (IL-6), Interleukin-6 (IL-8), and Tumor Necrosis Factor-alpha (TNF-alpha) to estimate systemic inflammatory response. Two sets of preoperative blood draws will be obtained. The first set (preoperative) will be drawn following consent during consultation. The second set (immediate preoperative) will be drawn just prior to the operation on Day 0. Participants will return to the office on postoperative day five (POD5) to have blood drawn for the third set of blood draws (postoperative). Concentrations for each of the inflammatory cytokines (IL-6, IL-8, and TNF- alpha) will be reported in pg/mL and results at each timepoint will be summarized by study arm using basic descriptive statistics.
Inflammatory markers - CRP concentrations | Blood draws during consultation, immediately prior to surgery, and at POD5, approximately 2-4 weeks total
  Preoperative and postoperative blood draws will be taken to measure concentrations of C-reactive protein (CRP). CRP is produced by the liver in response to pro-inflammatory cytokines released during inflammation. Two sets of preoperative blood draws will be obtained. The first set (preoperative) will be drawn following consent during consultation. The second set (immediate preoperative) will be drawn just prior to the operation on Day 0. Participants will return to the office on postoperative day five (POD5) to have blood drawn for the third set of blood draws (postoperative). CRP concentration will be reported in mg/L and results at each timepoint will be summarized by study arm using basic descriptive statistics.
Preoperative Anxiety | On the day of surgery prior to the procedure, approximately 2-4 weeks after enrollment
  Preoperative anxiety will be assessed using an Anxiolysis Questionnaire modeled on the Amsterdam Preoperative Anxiety and Information Scale (APAIS). Participants will complete the survey to describe anxiety levels immediately before surgery. This survey consists of 4 questions which asks participants to rate each item on a scale of 1 ("Not at all") to 5 ("Extremely" or "Extremely highly") to best describe how worried they are about the procedure and anesthetic as well as how often they think about the procedure and anesthetic. Higher scores are associated with increasing levels of anxiety with a total score of >=11 considered a key anxiety threshold. Scores will be summarized and reported using basic descriptive statistics.
Preoperative Sleep Quality | On the day of surgery prior to the procedure, approximately 2-4 weeks after enrollment
  Sleep quality over the previous three nights while taking the premedication immediately before surgery will be assessed based on a survey response. Specifically, participants will be administered a survey and asked to rate their quality of sleep during the three nights prior to surgery on a scale of 1 ("Much improved") to 5 ("Much worse") such that lower scores are associated with increased sleep quality. Sleep quality results will be presented as frequencies (percentages).
Post operative pain | The morning of the first 3 postoperative days (approximately 72 hours postoperatively) and during the postoperative appointment on POD 5, approximately 2-4 weeks.
  Post operative pain will be assessed using a Visual Analog Scale (VAS). The VAS is a unidimensional tool for measuring pain intensity. Participants will be administered a total of four surveys via text message or email with a link to SurveyMonkey. These surveys will be sent approximately 1 day, 2 days, and 3 days following surgery and will take about 2 minutes to complete. The last survey will be administered on paper during postoperative follow up, on POD5. The surveys will query for participant ID and then ask participants to describe the worst pain they have experienced since the surgery or since the previous survey depending on day administered, using the VAS. Responses for the VAS can range from 0-100 wherein 0 = "No pain" and 100 = "Worst pain imaginable" such that higher scores are indicative of greater pain intensity. Cut points on the VAS include "Mild" (1-30), "Moderate" (31-70) and "Severe" (71-100). Pain scores will be summarized using basic descriptive statistics.
Heart Rate | During consultation and again immediately preoperatively on the day of surgery, approximately 2-4 weeks total
  Heart rate will be measured twice during the study, once at the time of consultation and a second time immediately prior to surgery. Heart rate will be recorded in beats per minute (bpm) and summarized by study arm using basic descriptive statistics.
Mean Arterial Pressure (MAP) | During consultation and again immediately preoperatively on the day of surgery, approximately 2-4 weeks total
  Mean arterial pressure will be measured twice during the study, once at the time of consultation and a second time immediately prior to surgery. MAP will be recorded in millimeters of mercury (mmHg) and summarized by study arm using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Baker, DMD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center Department of Dentistry, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Background] Jones CM. Heroin use and heroin use risk behaviors among nonmedical users of prescription opioid pain relievers - United States, 2002-2004 and 2008-2010. Drug Alcohol Depend. 2013 Sep 1;132(1-2):95-100. doi: 10.1016/j.drugalcdep.2013.01.007. Epub 2013 Feb 12. PMID 23410617
- [Background] Cicero TJ, Ellis MS, Surratt HL, Kurtz SP. The changing face of heroin use in the United States: a retrospective analysis of the past 50 years. JAMA Psychiatry. 2014 Jul 1;71(7):821-6. doi: 10.1001/jamapsychiatry.2014.366. PMID 24871348
- [Background] Nasr, D. A., & Abdellatif, A. A. (2014). Efficacy of preoperative melatonin versus pregabalin on perioperative anxiety and postoperative pain in gynecological surgeries. Egyptian Journal of Anaesthesia, 30(1), 89-93. doi:10.1016/j.egja.2013.10.001
- [Background] Andersen LP, Werner MU, Rosenberg J, Gogenur I. A systematic review of peri-operative melatonin. Anaesthesia. 2014 Oct;69(10):1163-71. doi: 10.1111/anae.12717. Epub 2014 May 19. PMID 24835540
- [Background] Favero G, Franceschetti L, Bonomini F, Rodella LF, Rezzani R. Melatonin as an Anti-Inflammatory Agent Modulating Inflammasome Activation. Int J Endocrinol. 2017;2017:1835195. doi: 10.1155/2017/1835195. Epub 2017 Oct 1. PMID 29104591
- [Background] Ambriz-Tututi M, Rocha-Gonzalez HI, Cruz SL, Granados-Soto V. Melatonin: a hormone that modulates pain. Life Sci. 2009 Apr 10;84(15-16):489-98. doi: 10.1016/j.lfs.2009.01.024. Epub 2009 Feb 15. PMID 19223003
- [Background] de Carvalho Nogueira EF, de Oliveira Vasconcelos R, Teixeira Correia SS, Souza Catunda I, Amorim JA, do Egito Cavalcanti Vasconcelos B. Is There a Benefit to the Use of Melatonin in Preoperative Zygomatic Fractures? J Oral Maxillofac Surg. 2019 Oct;77(10):2017.e1-2017.e7. doi: 10.1016/j.joms.2019.05.016. Epub 2019 Jun 4. PMID 31260676
- [Background] Moerman N, van Dam FS, Muller MJ, Oosting H. The Amsterdam Preoperative Anxiety and Information Scale (APAIS). Anesth Analg. 1996 Mar;82(3):445-51. doi: 10.1097/00000539-199603000-00002. PMID 8623940
- [Background] Myles PS, Myles DB, Galagher W, Boyd D, Chew C, MacDonald N, Dennis A. Measuring acute postoperative pain using the visual analog scale: the minimal clinically important difference and patient acceptable symptom state. Br J Anaesth. 2017 Mar 1;118(3):424-429. doi: 10.1093/bja/aew466. PMID 28186223
- [Background] Viswanath A, Oreadi D, Finkelman M, Klein G, Papageorge M. Does Pre-Emptive Administration of Intravenous Ibuprofen (Caldolor) or Intravenous Acetaminophen (Ofirmev) Reduce Postoperative Pain and Subsequent Narcotic Consumption After Third Molar Surgery? J Oral Maxillofac Surg. 2019 Feb;77(2):262-270. doi: 10.1016/j.joms.2018.09.010. Epub 2018 Sep 20. PMID 30321520